CLINICAL TRIAL: NCT04313556
Title: Clinical Outcome of Arthroscopic Lateral Release for Lateral Patellar Compression Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Sherwan Ahmed Ali Hamawandi, Assistant professor of orthopedic surgery, Hawler Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMU/Sherwan8
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Knee Pain Chronic
Keywords: Lateral patellar compression syndrome; Arthroscopic lateral release; Lysholm score

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lateral patellar release (Other): Arthroscopic lateral patellar retinacular release
  Interventions: Procedure: Lateral patellar release

INTERVENTIONS:
Procedure: Lateral patellar release — Arthroscopic lateral patellar reticular release

SUMMARY:
We performed a prospective case series study of 48 patients who suffered Lateral patellar compression syndrome who were diagnosed by clinical examination and confirmed by M.R.I. and failed conservative management and underwent isolated arthroscopic lateral patellar retinaculum release in Erbil Teaching Hospital, PAR Private Hospital and Hawler Private Hospital between December 2016 and August 2019.

ELIGIBILITY:
Inclusion Criteria:

* Lateral patellar compression syndrome proved by clinical,MRI and Arthroscopic examination

Exclusion Criteria:

1. Dislocated or history of dislocation.
2. Patellar instability.
3. Bony abnormality (trochlear groove hypoplasia or flat).
4. Osteoarthritis of the knee 3rd and 4th grades.
5. Infected knee.
6. Varus and valgus knee.
7. Rotational deformity of the lower extremity.
8. Miserable malalignment triad.
9. Anterior cruciate ligament, posterior cruciate ligament and medial collateral ligament rupture.
10. History of fracture around knee.
11. Focal Osteoarthritis of the lateral facet joint.
12. Chondral lesion (Outerbridge 3 and 4).

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-12-04 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Lysholm Knee Score | 12 months
  Eight sections are assessed to produce an overall score on a scale of 0 to 100. Then an assignment is given as "excellent" for 95 to 100 points; "good" for 85 to 94 points, "fair" for 65 to 84 points, or "poor" for less than 65 points

IPD SHARING:
Plan to Share IPD: No